CLINICAL TRIAL: NCT05443178
Title: Open Label, Single Center, Phase 1 Dose Escalation and Extension Trial to Evaluate Safety and Tolerability of Chlorquine as Adjuvant Drug to Standard 4-drug Anti-tuberculosis Therapy in Healthy Volunteers
Brief Title: Safety and Tolerability of Chlorquine in Addition to Anti-tuberculosis Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Clear TB
Record Dates: First submitted 2020-08-20; First posted 2022-07-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Tuberculosis Infection
Keywords: Safety and tolerability; Chloroquin as adjuvant to standard 4-drug anti-TB therapy; Healthy volunteers; Phase I trial
MeSH Terms: conditions — Latent Tuberculosis | interventions — Chloroquine; Rifampin; Isoniazid; Ethambutol; Pyrazinamide

STUDY DESIGN:
Intervention Model Description: 3 subjects are planned to enter each cohort. No more than 3 subjects will receive the same dose during the dose escalation phase.
  3 participants are initially enrolled into the first dose cohort (100mg daily). If there is no DLT observed at Day 30, the investigators enroll 3 additional subjects into the second dose cohort (200mg daily). The targeted maximum dose of Nivaquine® is 300mg (cohort 3).
  Development of DLTs in ≥ 1 subject(s) in a specific dose cohort suggests that the RP2D has been exceeded, and further dose escalation is not pursued. In this case, the preceding dose level will be assumed to be the dose level for another 7 participants in the extension part of the study. If in cohort 3, no DLT is observed, an additional 7 participants will receive 300 mg chloroquine daily in the dose extension phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 100 mg Nivaquine and 4 Tabl Rimstar peroral once daily before breakfast for 14 days
  Interventions: Drug: Nivaquine ® (Chloroquine)
- Cohort 2 (Experimental): 200 mg Chloroquine and 4 Tabl Rimstar peroral once daily before breakfast for 14 days
  Interventions: Drug: Nivaquine ® (Chloroquine)
- Cohort 3 (Experimental): 300 mg Chloroquine and 4 Tabl Rimstar peroral once daily before breakfast for 14 days
  Interventions: Drug: Nivaquine ® (Chloroquine)
- Dose extension group (Experimental): Dose escalation: XX mg Chloroquine (depending on results) and 4 Tabl Rimstar peroral once daily before breakfast for 14 days
  Interventions: Drug: Nivaquine ® (Chloroquine)

INTERVENTIONS:
Drug: Nivaquine ® (Chloroquine) — dose escalation and extension trial
  Other Names: Rimstar ® (Rifampicin, Isoniazid, Ethambutol, Pyrazinamid)

SUMMARY:
In vitro and in vivo data show promising results of adjunctive use of Chloroquine to standard tuberculosis therapy as Chloroquine enhances animicrobial effectiveness against intracellular MTB. To date, no safety data of the concurrent use of both treatments is availble. In a phase I trial, the investigators aim to evaluate safety and tolerability of the concurrent use of Chloroquine and standard anti-TB drug in healthy volunteers.

DETAILED DESCRIPTION:
Even though tuberculosis (TB) remains one of the top 10 causes of death worldwide in 2019, there exists a gap in development of new diagnostics and treatments. There is a substantial need for new TB regimens, which would ideally be shorter, more tolerable and more efficient in eradicating all subpopulations of mycobacterium tuberculosis (MTB). In this regard, a promising TB drug pipeline emerges through re-use of marketed non TB-drugs, re-engineering of existing anti-TB compounds and discovery of new compounds. In vitro data showed that Chloroquine (CQ) inhibits an efflux pump expressed on macrophages. Inhibition of this pump increases intracellular concentration of Isoniazid and Pyrazinamide and enhances antimicrobial effectiveness against intracellular MTB. Recently published in vivo mouse model data confirmed the positive effect of CQ combined with the standard anti-TB therapy.

In line with global attempts to enhance effectiveness and shorten TB therapy, the investigators propose to evaluate this combination in a clinical setting. The absence of clinical study data showing safety and tolerability of CQ administered with first-line anti-TB drugs in humans shows the need for the research team to conduct this study. the investigators hypothesize that additional CQ to standard 4-drug anti-TB therapy is safe and increases the efficacy against intracellular MTB, leading to a pronounced reduction of the intracellularly hiding bacteria and overall to an accelerated reduction of bacterial load. The major advantages of this new combination with CQ and the 4-drug anti-TB therapy are, that all substances are long-term approved, commercially available drugs and that effective CQ concentrations are well achievable in humans.

Primary objective of the study is to investigate the safety and tolerability of a combination of standard doses of Nivaquine® (Chloroquine) with standard doses of Rimstar® (4-drug anti-TB therapy) in healthy volunteers.

Secondary objective of the study is to assess drug concentration of the new combination (Nivaquine® and Rimstar®) in healthy volunteers over time.

ELIGIBILITY:
Inclusion criteria:

1. Informed study-specific consent (including possible pharmacogenetic analysis) as documented by signature
2. Healthy volunteers aged between 18 and 50 years of age (significantly increased risk of side effects from 50 years of age with Rimstar®)

Exclusion criteria:

1. Lack of highly effective contraception during the study treatment and for 8 months after the last dose of study treatment (until Day 254, visit 7) according to 11.4 with the following consideration for participating women:

   * From Day 1 (visit 2) up to Day 30 (visit 6) hormonal contraception is insufficient due to lower concentrations of estrogen and/or gestagen during and up to 14 days after Rimstar® intake. The hormonal contraception must be supplemented with a barrier method (preferably male condom).
   * From Day 30 (visit 6) up to Day 254 (visit 7) hormonal contraceptive methods can be used and are considered highly effective.
2. Pregnant or lactating females
3. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product, glucose-6-phosphate dehydrogenase insufficiency (favism)
4. Regular treatment with drugs in the last 14 days prior to first intake of study drug (except for Paracetamol and Vitamin B6 (pyridoxine), see 8.7).
5. History of or concurrent, clinically significant cardiac, immunological, pulmonary, neurological, renal, gastrointestinal, dermatological, endocrinological or other major disease as determined by the Investigator and/or his representative
6. History of or presence of any clinically significant abnormality in vital signs, ECG, or laboratory test results or has any medical or psychiatric condition that, in the opinion of the Investigator, may interfere with the study procedures or compromise subject safety
7. History of or currently present retinopathy or other disturbances of the field of vision or the retina according to the Investigator
8. History of alcohol or substance abuse for the last 3 months prior to Screening, as determined by the Investigator
9. Weight less than 55kg
10. Intake of grapefruit juice or grapefruits within 2 weeks before the first study drug administration and during treatment phase
11. Donation of blood or blood products within a 30-day period prior to Screening
12. Current enrolment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 3 months of participation to the Clear trial.
13. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
14. The investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-10-04 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Physicial examination 1.1 | day 14
  Heart auscultation (normal/abnormal)
Physicial examination 1.2 | day 30
  Heart auscultation (normal/abnormal)
Physicial examination 2.1 | day 14
  lung auscultation (normal, abnormal)
Physicial examination 2.2 | day 30
  lung auscultation (normal, abnormal)
Physicial examination 3.1 | day 14
  abdominal examination (normal, abnormal)
Physicial examination 3.2 | day 30
  abdominal examination (normal, abnormal)
Physicial examination 4.1 | day 14
  lymph node palpation (normal, abnormal)
Physicial examination 4.2 | day 30
  lymph node palpation (normal, abnormal)
Physicial examination 5.1 | day 14
  reflex testing (normal, abnormal)
Physicial examination 5.2 | day 30
  reflex testing (normal, abnormal)
Physicial examination 6.1 | day 14
  test vibration sense with tuning fork (mallelor left and right X/8)
Physicial examination 6.2 | day 30
  test vibration sense with tuning fork (mallelor left and right X/8)
Vital Signs 1.1 | day 1
  heart rate (beats/min)
Vital Signs 1.2 | day 7
  heart rate (beats/min)
Vital Signs 1.3 | day 14
  heart rate (beats/min)
Vital Signs 1.4 | day 15
  heart rate (beats/min)
Vital Signs 1.5 | day 30
  heart rate (beats/min)
Vital Signs 2.1 | day 1
  blood pressure (mmHg)
Vital Signs 2.2 | day 7
  blood pressure (mmHg)
Vital Signs 2.3 | day 14
  blood pressure (mmHg)
Vital Signs 2.4 | day 15
  blood pressure (mmHg)
Vital Signs 2.5 | day 30
  blood pressure (mmHg)
Vital Signs 3.1 | day 1
  temperature (°C)
Vital Signs 3.2 | day 7
  temperature (°C)
Vital Signs 3.3 | day 14
  temperature (°C)
Vital Signs 3.4 | day 15
  temperature (°C)
Vital Signs 3.5 | day 30
  temperature (°C)
Safety Laboratory samples Panel 1.1 | day 1
  Sodium (mmol/l)
Safety Laboratory samples Panel 1.2 | day 7
  Sodium (mmol/l)
Safety Laboratory samples Panel 1.3 | day 14
  Sodium (mmol/l)
Safety Laboratory samples Panel 1.4 | day 30
  Sodium (mmol/l)
Safety Laboratory samples Panel 2.1 | day 1
  Potassium (mmol/l)
Safety Laboratory samples Panel 2.2 | day 7
  Potassium (mmol/l)
Safety Laboratory samples Panel 2.3 | day 14
  Potassium (mmol/l)
Safety Laboratory samples Panel 2.4 | day 30
  Potassium (mmol/l)
Safety Laboratory samples Panel 3.1 | day 1
  Calcium (mmol/l)
Safety Laboratory samples Panel 3.2 | day 7
  Calcium (mmol/l)
Safety Laboratory samples Panel 3.3 | day 14
  Calcium (mmol/l)
Safety Laboratory samples Panel 3.4 | day 30
  Calcium (mmol/l)
Safety Laboratory samples Panel 4.1 | day 1
  Creatinine (umol/l)
Safety Laboratory samples Panel 4.2 | day 7
  Creatinine (umol/l)
Safety Laboratory samples Panel 4.3 | day 14
  Creatinine (umol/l)
Safety Laboratory samples Panel 4.4 | day 30
  Creatinine (umol/l)
Safety Laboratory samples Panel 5.1 | day 1
  Total Bilirubin (umol/l)
Safety Laboratory samples Panel 5.2 | day 7
  Total Bilirubin (umol/l)
Safety Laboratory samples Panel 5.3 | day 14
  Total Bilirubin (umol/l)
Safety Laboratory samples Panel 5.4 | day 30
  Total Bilirubin (umol/l)
Safety Laboratory samples Panel 6.1 | day 1
  ALT (U/l)
Safety Laboratory samples Panel 6.2 | day 7
  ALT (U/l)
Safety Laboratory samples Panel 6.3 | day 14
  ALT (U/l)
Safety Laboratory samples Panel 6.4 | day 30
  ALT (U/l)
Safety Laboratory samples Panel 7.1 | day 1
  Glucose (mmol/l)
Safety Laboratory samples Panel 7.2 | day 7
  Glucose (mmol/l)
Safety Laboratory samples Panel 7.3 | day 14
  Glucose (mmol/l)
Safety Laboratory samples Panel 7.4 | day 30
  Glucose (mmol/l)
Safety Laboratory samples Panel 8.1 | day 1
  CRP (mg/l)
Safety Laboratory samples Panel 8.2 | day 7
  CRP (mg/l)
Safety Laboratory samples Panel 8.3 | day 14
  CRP (mg/l)
Safety Laboratory samples Panel 8.4 | day 30
  CRP (mg/l)
Safety Laboratory samples Panel 9.1 | day 1
  Haemoglobin (g/l)
Safety Laboratory samples Panel 9.2 | day 7
  Haemoglobin (g/l)
Safety Laboratory samples Panel 9.3 | day 14
  Haemoglobin (g/l)
Safety Laboratory samples Panel 9.4 | day 30
  Haemoglobin (g/l)
Safety Laboratory samples Panel 10.1 | day 1
  Platlets (G/l)
Safety Laboratory samples Panel 10.2 | day 7
  Platlets (G/l)
Safety Laboratory samples Panel 10.3 | day 14
  Platlets (G/l)
Safety Laboratory samples Panel 10.4 | day 30
  Platlets (G/l)
Safety Laboratory samples Panel 11.1 | day 1
  White blood cell (G/l)
Safety Laboratory samples Panel 11.2 | day 7
  White blood cell (G/l)
Safety Laboratory samples Panel 11.3 | day 14
  White blood cell (G/l)
Safety Laboratory samples Panel 11.4 | day 30
  White blood cell (G/l)
Safety Laboratory samples Panel 12.1 | day 7
  Blood pregnancy test (Blood beta-hCG)
Safety Laboratory samples Panel 12.2 | day 30
  Blood pregnancy test (Blood beta-hCG)
Urinanalysis 1.1 | day 1
  Dipstick: protein negative/+/++/+++
Urinanalysis 1.2 | day 7
  Dipstick: protein negative/+/++/+++
Urinanalysis 1.3 | day 14
  Dipstick: protein negative/+/++/+++
Urinanalysis 1.4 | day 30
  Dipstick: protein negative/+/++/+++
Urinanalysis 2.1 | day 1
  Dipstick: white blood cells negative/+/++/+++
Urinanalysis 2.2 | day 7
  Dipstick: white blood cells negative/+/++/+++
Urinanalysis 2.3 | day 14
  Dipstick: white blood cells negative/+/++/+++
Urinanalysis 2.4 | day 30
  Dipstick: white blood cells negative/+/++/+++
Urinanalysis 3.1 | day 1
  Dipstick: red blood cells negative/+/++/+++
Urinanalysis 3.2 | day 7
  Dipstick: red blood cells negative/+/++/+++
Urinanalysis 3.3 | day 14
  Dipstick: red blood cells negative/+/++/+++
Urinanalysis 3.4 | day 30
  Dipstick: red blood cells negative/+/++/+++
Urinanalysis 4.1 | day 1
  Dipstick: Glucose negative/+/++/+++
Urinanalysis 4.2 | day 7
  Dipstick: Glucose negative/+/++/+++
Urinanalysis 4.3 | day 14
  Dipstick: Glucose negative/+/++/+++
Urinanalysis 4.4 | day 30
  Dipstick: Glucose negative/+/++/+++
Safety 12 lead ECG 1.1 | day 7
  Rate/min
Safety 12 lead ECG 1.2 | 30
  Rate/min
Safety 12 lead ECG 2.1 | day 7
  Rhythm (regular/irregular)
Safety 12 lead ECG 2.2 | day 30
  Rhythm (regular/irregular)
Safety 12 lead ECG 3.1 | day 7
  PQ interval (ms)
Safety 12 lead ECG 3.3 | day 30
  PQ interval (ms)
Safety 12 lead ECG 4.1 | day 7
  QRS interval (ms)
Safety 12 lead ECG 4.2 | day 30
  QRS interval (ms)
Safety 12 lead ECG 5.1 | day 7
  ST Segment (normal/elevation/depression)
Safety 12 lead ECG 5.2 | day 30
  ST Segment (normal/elevation/depression)
Safety ophtalmological examination 1.1 | day 30
  Slit lamp examaniation both sides (normal/abnormal)
Safety ophtalmological examination 1.2 | day 30
  Refraction both sides (+/-)
Safety ophtalmological examination 1.3 | day 30
  Biomicroscopy of the central fundus both sides(normal/abnormal)
Safety ophtalmological examination 1.4 | day 30
  Applanation tonometry and stereoscopic papilla evaluation bilateral (normal/abnormal), Color sense test according to Panel D-15 right and left side (normal/abnormal)
Safety ophtalmological examination 1.5 | day 30
  Color sense test according to Panel D-15 bilateral (normal/abnormal)
Occurence of adverse events and serious adverse events 1.1 | day 1
  according to GCP Guideline
Occurence of adverse events and serious adverse events 1.2 | day 7
  according to GCP Guideline
Occurence of adverse events and serious adverse events 1.3 | day 14
  according to GCP Guideline
Occurence of adverse events and serious adverse events 1.4 | day 15
  according to GCP Guideline
Occurence of adverse events and serious adverse events 1.5 | day 30
  according to GCP Guideline
Occurence of adverse events and serious adverse events 1.6 | day 256
  according to GCP Guideline

SECONDARY OUTCOMES:
Drug concentration over time measured by the pharmacokinetics | day 14 prior to dosing (-15 until -5 minutes) and 1, 2, 4, 6 and 24 hours after dosing
  drug concentration (mg/l) of Rifampicin, Isoniazid, 25-O-Desacetylrifampicin, Ethambutol, Pyrazinamide, Chloroquine, Desethylchloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Kaelin, Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Clinical Trial Center, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No